CLINICAL TRIAL: NCT07378007
Title: Body Composition and Characteristics of Performance in Collegiate Cheerleaders and Dancers
Brief Title: Characteristics of Performance in Collegiate Cheerleaders and Dancers
Status: Recruiting | Type: Observational
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Director, FSU Institute of Sports Sciences and Medicine, Florida State University
Other Study IDs: CDNWO00006460
Record Dates: First submitted 2026-01-14; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Low Energy Availability; Physical Performance; Nutrition
Keywords: Body Composition; Energy Availability; Physical Fitness; Division I Collegiate Cheerleaders and Dancers; Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Division I Collegiate Cheerleaders and Dancers: Normal weight obese or normal weight lean

SUMMARY:
This study aims to investigate performance differences between collegiate cheerleaders and dancers classified as normal weight obese and those classified as normal weight lean. The study will assess differences in physical performance, lifestyle behaviors, muscle quality, and nutrition-related factors between groups. Performance testing, body composition assessment, and questionnaire-based measures will be used to characterize these relationships.

DETAILED DESCRIPTION:
This study focuses on understanding body composition-related differences in performance among collegiate cheerleaders and dancers, a population that relies heavily on strength, power, and aesthetic presentation for successful performance. Obesity is commonly classified using body mass index (BMI); however, BMI may fail to identify individuals with excess adiposity, particularly in athletic populations. One such classification is normal-weight obesity, which describes individuals with a normal BMI but elevated body fat percentage and increased risk for impaired muscle function and reduced physical performance. Aesthetic athletes, including cheerleaders and dancers, may be particularly susceptible to this condition due to sport-specific performance demands and body composition expectations. This study aims to determine whether performance outcomes differ between normal weight obese and normal weight lean cheerleaders and dancers, with specific focus on measures of power, strength, and muscle quality. In addition, the study examines differences in lifestyle behaviors, compositional and functional muscle characteristics of the upper leg, and nutrition-related factors between groups. By integrating body composition assessment, physical performance testing, and questionnaire-based measures, this study seeks to better characterize normal-weight obesity in this population. Ultimately, the findings may help clarify how body composition and lifestyle factors relate to performance in collegiate cheer and dance athletes.

ELIGIBILITY:
Inclusion Criteria:

* Must be a part of either the Florida State University dance or cheer team
* Sex: Female
* Age: 18-30
* BMI: Normal (18.5 - 24.9 kg/m2)

Exclusion Criteria:

* Not biologically female
* Have a diagnosed and unresolved eating disorder
* Not weight stable (defined as a gain/loss of more than ~7.7 lbs in the past 2 months)
* Participants who are pregnant or who become pregnant during the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Current members of the Florida State University Cheer and Dance teams
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2025-08-03 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Energy Availability (kcals/kg FFM) | 7 days
  Energy availability will be assess by subtracting exercise energy expenditure from energy intake relative to fat free mass. This will be assessed daily for 7 continuous days.
Physical Fitness | Day of study enrollment
  Physical fitness will be assessed via maximal jump height (in inches) using a double leg (and single leg counter movement jump and a maximal isokinetic leg extension and leg curl (expressed in kgs).

SECONDARY OUTCOMES:
Subjective Sleep | Day of study enrollment
  The Pittsburgh Sleep Quality Index (PSQI) will be used to assess subjective sleep quality, while the Athlete Sleep Behavior Questionnaire (ASBQ) will be used to assess subjective sleep behavior. A score of >42 on the ASBQ indicates poor sleep behavior. A score >5 on the PSQI indicates poor sleep quality.
Body Composition | Day of study enrollment
  Body Composition will be assessed via Air Displacement Plethysmography on the first day of study enrollment.
Muscle Quality - Echo Intensity | Day of study enrollment
  Ultrasound echo intensity will be used to assess intramuscular fat.
Nutrition Knowledge | Day of study enrollment
  Knowledge of nutrition based on the Abbreviated Nutrition for Sports Knowledge Questionnaire (ANSKQ). The maximum score is 100%. The minimum score is 0%. Higher scores indicate better nutrition knowledge.
Muscle Quality - Muscle Thickness | day of study enrollment
  Muscle thickness of the rectus femoris will be assessed via ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Sciences and Medicine (ISSM), Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided